CLINICAL TRIAL: NCT06157528
Title: Diagnosis of Pelvic Endometriosis: a Preliminary Study on the Added Value of R2*MFGRE Sequence in MRI
Brief Title: Diagnosis of Pelvic Endometriosis in MRI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhenshen Ma (Other)
Responsible Party: Sponsor-Investigator, Zhenshen Ma, Professor, Qianfoshan Hospital
Organization: Qianfoshan Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1110000
Record Dates: First submitted 2023-11-02; First posted 2023-12-06 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-12

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- ovarian endometriomas (Experimental): Patients received a single dose of 1OOmg abarelix injection with slow absorption, Cmax of (43.4±32.3)ng/mL, Tmax of (3.0±2.9) days. AUC0-∞ is (500 ±96) ng·d/mL, t1/2 is (13.2±3.2) days, CL/F is (208±48) L/d
  Interventions: Diagnostic Test: Magnetic resonance imaging

INTERVENTIONS:
Diagnostic Test: Magnetic resonance imaging — Patients were treated with abarelix prior to the examination

SUMMARY:
Purpose： Evaluate the feasibility of R2 star multiple fast gradient recalled echo (R2*MFGRE) imaging in the diagnosis of pelvic endometriosis.

One hundred patients with suspected endometriosis underwent routine pelvic MRI and R2*MFGRE imaging. Clinical diagnosis was pathologically confirmed one month after MRI examination. Three radiologists who were blinded to the pathological results evaluated the numbers of ovarian endometriomas (OMAs) and deep in-filtrating endometriosis (DIE) lesions using routine MRI and its combination with R2*MFGRE. MRI changes of lesion size before and after estrogen therapy.

DETAILED DESCRIPTION:
This prospective study was approved by the Ethics Committee of the local hos-pital, and informed consent was obtained from all the patients in this study (3701027061515). All procedures performed in studies involving human participants were in accordance with the ethical standards of our institutional and national re-search committee and with the Declaration of Helsinki.

Study population One hundred and Sixty-five patients with suspected endometriosis underwent pelvic MRI with R2*MFGRE imaging from Decemberr 2017 to December 2023. Of those, One hundred and forty patients were submitted to surgical (either laparotomy or laparoscopy) treatment for endometriosis. The diagnosis was confirmed by pathology within one month after the initial MR exam. Additionally, 20 out of 160 patients were excluded from the study. Of these, 11 were due to non-surgical treatment, and the other 8 were due to prominent susceptibility artifacts caused by colonic overdistention, limiting the vis-ibility of the pelvis. Finally, One hundred patients were included in the study.

All 100 patients were aged ranging from 24 to 54 years, with an average age of 37.8 years. Their clinical symptoms included dysmenorrhea, bulging in the lower abdomen or anus, heavy menstrual bleeding, dyspareunia, and infertility. Some of these patients had multiple symptoms

ELIGIBILITY:
Inclusion Criteria:

* patients who proven endometriosis by pathology Patients who wish to be treated

Exclusion Criteria:

* Received any treatment (radiotherapy, chemotherapy, surgery or chemoradiotherapy) before undergoing imaging studies poor-quality MR images with any severe motion or artifacts

Ages: 16 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Only women develop endometriosis
Enrollment: 100 (Estimated)
Dates: Start 2023-12-20 (Estimated); Primary Completion 2028-11 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Measuring the number of lesions | immediately after the surgery
  Pre- surgery, the number of lesions was counted during Magnetic resonance imaging by radiologists.
  Immediately after the intervention, the number of lesions found during the operation was counted by the surgeon.